CLINICAL TRIAL: NCT07084649
Title: The Efficacy of Dual-target iTBS in Youth With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Dual-target iTBS for Youth With ADHD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB, SMHC, 2025-01
Record Dates: First submitted 2025-07-04; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Phase 1 is an open-label, single-arm study to explore the preliminary efficacy, safety, and acceptability of aiTBS for youth with ADHD.
  • Phase 2 is a randomized, double-masked, controlled trial that will rigorously validate the results of Phase 1.
  The decision to proceed depends on Phase 1 results:
  * If Phase 1 demonstrates positive outcomes in clinical symptoms, cognitive functioning, safety, and acceptability, Phase 2 will be implemented.
  * If Phase 1 fails to show positive results, Phase 2 will be discontinued.
Masking Description: Phase 1：open label；Phase 2: double-blind masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1: Open-label dual-target aiTBS (Experimental): Phase 1: Open label, single arm study to determine the preliminary efficacy, safety, and acceptability of aiTBS for youth with ADHD.
  Interventions: Device: TMS
- Phase 2: RCT design active aiTBS (Active Comparator): Phase 1: A randomized, double-masked, controlled trial that will rigorously validate the efficacy and safety of dual-target aiTBS for youth with ADHD.
  Interventions: Device: TMS
- Phase 2: RCT design sham aiTBS (Sham Comparator): Phase 2: A randomized, double-masked, controlled trial that will rigorously validate the efficacy and safety of dual-target aiTBS for youth with ADHD.
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — accelerated intermittent theta burst stimulation

SUMMARY:
This study will employ accelerated intermittent theta burst stimulation (aiTBS) targeting two transcranial magnetic stimulation (TMS) sites: the right inferior frontal gyrus and left inferior parietal lobule.

DETAILED DESCRIPTION:
ADHD is the most common neurodevelopmental disorder in childhood. First-line clinical treatments primarily rely on psychostimulants, yet approximately 30% of adolescents with ADHD show inadequate response to current therapies. There is an urgent need to develop novel, practical, and sensitive intervention strategies.

Repetitive Transcranial Magnetic Stimulation (rTMS), a non-invasive technique that modulates neural activity via magnetic fields applied to brain regions beneath the skull, can induce long-lasting positive changes in neuroplasticity. This provides an alternative therapeutic approach for ADHD. In clinical research, rTMS has demonstrated potential value in treating children with ADHD. Notably, current studies have limitations: lack of control groups makes it difficult to exclude placebo effects, and the commonly used DLPFC target shows suboptimal efficacy in improving both clinical symptoms and cognitive functions, indicating room for improvement.

This study will be conducted in two phases:

* Phase 1 is an open-label, single-arm study to explore the preliminary efficacy, safety, and acceptability of aiTBS for youth with ADHD.
* Phase 2 is a randomized, double-masked, controlled trial that will rigorously validate the efficacy and safety of dual-target aiTBS and establish causal conclusions through a controlled design.

The decision to proceed depends on Phase 1 results:

* If Phase 1 demonstrates positive outcomes in clinical symptoms, cognitive functioning, safety, and acceptability, Phase 2 will be implemented.
* If Phase 1 fails to show positive results, Phase 2 will be discontinued.

The study will utilize MRI-guided neuronavigation to precisely locate the target brain regions (the right inferior frontal gyrus and the left inferior parietal lobule) for each participant. An aiTBS protocol will be employed. Based on a 90% resting motor threshold (adjusted for cortical depth), each participant will receive 10 iTBS sessions (1,800 pulses per session, with 60-minute inter-session intervals), administered twice daily over five consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. ADHD Diagnosis: Meets the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5);
2. Inadequate Response to Medication: After a full course of pharmacological treatment, the SNAP-IV Parent Rating Scale (first 18 items, assessing inattention/hyperactivity-impulsivity) score >1, and the Clinical Global Impression-Severity Scale (CGI-S) score >2;
3. Age and Gender: 10-18 years old; males or females;
4. Intellectual Functioning: Full-scale intelligence quotient (IQ) >70 on the China-Wechsler Intelligence Scale for Children (C-WISC) (excluding participants with intellectual disability);
5. Symptom Severity: A score of ≥1.6 on either the Inattention or Hyperactivity/Impulsivity subscale of the SNAP-IV Parent Rating Scale;
6. Medication Requirements:

1) Medication-naïve or currently off medication; 2) If currently on medication, must be on a stable medication regimen for at least 4 weeks prior to the baseline visit and throughout the study duration; 3) Prohibited medications: Psychostimulants; 7. Right-handed.

Exclusion Criteria:

1. Contraindications for TMS therapy include epilepsy, cardiac pacemakers, cochlear implants, and metal implants.
2. Contraindications for MRI include metal implants in the body, claustrophobia, and tattoos.
3. Significant medical history: history of epilepsy, organic brain disorders, traumatic brain injury (TBI), or severe physical illnesses.
4. Behavioral risks: history of violent or suicidal behavior.
5. Comorbid neurodevelopmental disorders, such as autism spectrum disorder (ASD), tic disorders, etc.
6. Comorbid psychiatric disorders: any other primary psychiatric disorders, except conduct disorder/oppositional defiant disorder, mild anxiety, or depression.
7. Substance abuse.
8. Currently receiving any non-medical treatments, such as cognitive behavioral therapy (CBT), neurofeedback, etc.
9. Female participants must not be pregnant or breastfeeding.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness as measured by SNAP-IV Parent Rating Scale (assessing inattention/hyperactivity-impulsivity) | ADHD symptoms will be measured before the TMS treatment, immediately after completion of the TMS treatment.
  SNAP-IV is used to assess the core symptoms of ADHD (inattention, hyperactivity/impulsivity) and symptoms of oppositional defiant disorder; the total score or subscale mean scores indicate symptom severity, with higher scores reflecting more pronounced symptoms.
Clinical Global Impression-Severity Scale (CGI) | GCI will be measured before the TMS treatment, immediately after completion of the TMS treatment.
  CGI is used to evaluate disease severity and treatment response.

SECONDARY OUTCOMES:
Safety as measured by number of participants with Adverse Events | Each afternoon after treatment during the 5 days of treatment
  Count of Adverse Events Reported during follow up
Acceptability as assessed by treatment-related dropout rates | Each afternoon after treatment during the 5 days of treatment
  Acceptability is assessed by treatment-related dropout rates, such as dropouts due to TMS side effects or lack of efficacy
BRIEF（Behavior Rating Inventory of Executive Function） | Will be measured before the TMS treatment, immediately after completion of the TMS treatment.
  To assess behavioral manifestations of executive function in children, and adolescents
PedsQL（Pediatric Quality of Life Inventory） | Will be measured before the TMS treatment, immediately after completion of the TMS treatment.
  To measure health-related quality of life in children and adolescents, covering physical, emotional, and social functioning.
A cognitive task battery | Will be measured before the TMS treatment, immediately after completion of the TMS treatment.
  Trail Making Test (TMT): Part A; WMS III Spatial Span; Brief Visuospatial Memory Test-Revised NAB Mazes; CPT-IP; N-back task; Go/No-Go task; Flanker tasks.
Cortical excitability and cortical inhibition function indicators | Will be measured before the TMS treatment, immediately after completion of the TMS treatment.
  Resting motor threshold, 1mV motor evoked potential threshold and amplitude, short-interval cortical inhibition and intracortical facilitation

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, None Selected, China

IPD SHARING:
Plan to Share IPD: No
This requires approval from our institution's ethics committee.